CLINICAL TRIAL: NCT01937624
Title: Pediatric Distal Radius US Study
Status: Completed | Type: Observational
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00021828
Record Dates: First submitted 2013-08-28; First posted 2013-09-09 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Distal Radius Fractures
Keywords: Diagnostic ultrasound
MeSH Terms: conditions — Wrist Fractures | interventions — Ultrasonography; X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic ultrasound and radiographic imaging: - The diagnostic musculoskeletal ultrasound and x-rays will both be used to image bones in perpendicular and orthogonal planes over the distal radius visualizing the physis.
  Interventions: Device: Diagnostic Ultrasound; Radiation: X-ray imaging

INTERVENTIONS:
Device: Diagnostic Ultrasound
  Other Names: Sonosite Ultrasound
Radiation: X-ray imaging

SUMMARY:
The purpose of the study is to evaluate the sensitivity and specificity of using a diagnostic musculoskeletal ultrasound in pediatric distal radius fractures in an outpatient setting. Ultrasound reliability and accuracy will be tested. The result of the diagnostic ultrasound will be compared to x-ray diagnosis under routine conditions in the investigator's injury and fracture treatment evening clinic. Data will be collected and recorded during the duration of the 12 week study. Through the literature review and experience with ultrasound, the investigators anticipate that diagnostic ultrasound will provide very high sensitivity and specificity in diagnosing distal radius fractures in children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient with a wrist injury.

Exclusion Criteria:

* Gross deformity of the injured body part, suspected open fractures and the need for emergent surgery

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with wrist injury
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Cassas, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Hospital System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas - Greenville Hospital System, Greenville, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic Ultrasound and Radiographic Imaging: The diagnostic musculoskeletal ultrasound and x-ray will both be used to image bones in perpendicular and orthogonal planes over the distal radius visualizing the physis.
  Diagnostic Ultrasound
Period: Overall Study
Arm/Group | Diagnostic Ultrasound and Radiographic Imaging
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Diagnostic Ultrasound and Radiographic Imaging: The diagnostic musculoskeletal ultrasound and x-ray will both be used to image bones in perpendicular and orthogonal planes over the distal radius visualizing the physis.
Arm/Group | Diagnostic Ultrasound and Radiographic Imaging
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 51
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Presence of Fracture
Description: Diagnostic ultrasound will be used to determine if the bones do or do not have a fracture. Fractures will be based on the presence or absence of cortical disruption or irregularity on the ultrasound.
Time Frame: Duration of office visit
Population: Each of the 51 participants received both an ultrasound and a x-ray.
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic Ultrasound and Radiographic Imaging
Number analyzed (Participants) | 51
Participants
  Ultrasound: Fracture YES | 35
  Ultrasound: Fracture No | 16
  X Ray: Fracture YES | 34
  X Ray: Fracture No | 17

ADVERSE EVENTS:
Time Frame: N/A (No follow-up)
Description: All patients were monitored during their participation in the data collection process for adverse event occurrences.
Arm/Group | Diagnostic Ultrasound and Radiographic Imaging
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No